CLINICAL TRIAL: NCT02317952
Title: A Double-Blind, Randomized, Crossover Allergy Study of an Experimental Formula Followed by a 16 Week Double Blind Feeding Period to Assess Growth, Safety and Development of Tolerance to Cow's Milk Protein
Brief Title: Formula for Children With Cow's Milk Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perrigo Nutritionals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: PRG-VA-14-001
Record Dates: First submitted 2014-12-02; First posted 2014-12-17 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Extensively Hydrolyzed Formula (Experimental): Administered in context of oral food challenge and then for 16 weeks.
  Interventions: Other: Experimental Extensively Hydrolyzed Formula
- Comparator Formula (Active Comparator): Administered in context of oral food challenge and then for 16 weeks.
  Interventions: Other: Active Comparator Formula

INTERVENTIONS:
Other: Experimental Extensively Hydrolyzed Formula
  Arms: New Extensively Hydrolyzed Formula
Other: Active Comparator Formula
  Arms: Comparator Formula

SUMMARY:
The purpose of this study is to determine if a new extensively hydrolyzed formula can be consumed by children with Cow's Milk Allergy.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Parent/guardian must be willing to provide informed consent
* Parent/guardian agrees to feed study formula provided
* Confirmation of Cow's Milk Allergy

Exclusion Criteria:

* No clinically significant abnormal findings on medical history, laboratory results, and physical exam.
* No medications that may interfere with or impact evaluation of the study assessments
* Allergy to extensively hydrolyzed casein formula
* Tolerance of 200 ml of cow's milk, cow's milk-based formula or food products containing intact cow's milk protein within 2 weeks of the Screening Visit
* Participation in another clinical trial within 30 days of screening where they are are receiving an active intervention

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Allergic Reaction | 2 weeks

SECONDARY OUTCOMES:
Growth | 16 weeks
  Anthropometric measurements of weight in all enrolled subjects.
Growth | 16 weeks
  Anthropometric measurements of length/height in all enrolled subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy M Barber, PhD, Study Director — Perrigo Nutritionals
Locations (18):
- United States (18):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Arkansas Children's Hosptial, Little Rock, Arkansas
  - Pediatric Care Medical Group, Huntington Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Choc Psf, Amc, Orange, California
  - Allergy Medical Group of the North Area, INC, Roseville, California
  - Allergy & Asthma Medical Group and Research Center, APC, San Diego, California
  - 1st Allergy and Clinical Research Group, INC, d/b/a IMMUNOe International Research Centers, Centennial, Colorado
  - Sneeze Wheeze and Itch Associates, Normal, Illinois
  - Institute for Allergy and Asthma, Chevy Chase, Maryland
  - Einstein Consulting Services, LLC & Virgo Carter Pediatrics, Silver Spring, Maryland
  - Clinical Research Institute, Plymouth, Minnesota
  - Clinical Research Solutions, LLC, Middleburg Heights, Ohio
  - Allergy, Asthma, and Clinical Research Center, Oklahoma City, Oklahoma
  - Carolina Ear Nose and Throat Clinic, Orangeburg, South Carolina
  - TTS Research, Boerne, Texas
  - STAAMP Clinical Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington